CLINICAL TRIAL: NCT00205790
Title: Comparison of Primary Patency Between GORE-TEX PROPATEN Vascular Grafts and Thin Walled GORE-TEX Stretch Vascular Grafts
Brief Title: GORE-TEX PROPATEN Vascular Graft Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPT-01-04
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2008-08

CONDITIONS: Peripheral Vascular Diseases
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Vascular Grafting

INTERVENTIONS:
Device: Vascular graft

SUMMARY:
To demonstrate equivalence in patency performance of GORE-TEX PROPATEN Vascular Grafts and Thin Walled GORE-TEX Stretch Vascular Grafts in a peripheral bypass application to support a claim of substantial equivalence.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires primary above-knee bypass where the proximal anastomosis will be to the common femoral or proximal superficial femoral artery and the distal anastomosis will be the popliteal artery proximal to the medial head of the gastrocnemius;
* Patient has Grade III or IV occlusive vascular disease;
* Patient has a postoperative life expectancy greater than one year;
* Patient is at least 21 years of age;
* Patient is able to comply with all study requirements and be available for follow-up visits at 1 month, 6 months and 12 months post procedure;
* Patient is willing and able to provide written, informed consent.

Exclusion Criteria:

* Patient had a previous bypass in the diseased extremity (below iliacs);
* Patient has known coagulation disorders including hypercoagulability;
* Patient has had any previous instance of Heparin Induced Thrombocytopenia type 2 (HIT-2) or has known hypersensitivity to heparin;
* Patient has an acute embolic arterial occlusion;
* Patient requires sequential extremity revascularizations or other procedures that require use of additional vascular grafts;
* Patient had percutaneous transluminal angioplasty to the implant site within the previous 30 days;
* Patient is in need of, or is scheduled for, a cardiac surgical procedure or a different vascular surgical procedure;
* Patient has active infection in the region of graft placement; or
* Patient has an incomplete preoperative assessment (as outlined in this protocol) due to an emergency procedure, a traumatic injury or any other reason.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2003-02; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Primary patency at 12 months
Major device complication rates at 12 months

SECONDARY OUTCOMES:
Technical failures
Secondary patency

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Ascher, MD, Principal Investigator — Maimonides Hospital, Brooklyn NY
Locations (18):
- United States (18):
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Memorial Regional Hospital, Hollywood, Florida
  - St. Vincent's Hospital, Jacksonville, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Medical Center of Central Georgia, Macon, Georgia
  - Jewish Hospital, Louisville, Kentucky
  - Upper Chesapeake Medical Center, Baltimore, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - William Beaumont Hospital, Bingham Farms, Michigan
  - Borgess Hospital, Kalamazoo, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Maimonides Hospital, Brooklyn, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - Wilkes-Barre General Hospital, Plains, Pennsylvania
  - Baptist East Hospital, Memphis, Tennessee
  - Charleston Area Medical Center, Charleston, West Virginia